CLINICAL TRIAL: NCT03246256
Title: Recall of Information on Intravenous Thrombolysis in Acute Ischaemic Stroke Patients Given During Informed Consent: a Prospective Observational Study.
Brief Title: Information Recall on Informed Consent to Intravenous Thrombolysis in Patients With Acute Ischaemic Stroke.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Department of Neurology, Charité - Universitätsmedizin Berlin, Germany (Unknown); Department of Cardiology and Pneumology, Charité, Campus Benjamin Franklin (Unknown)
Responsible Party: Principal Investigator, Karl Georg Haeusler, Consultant Neurologist, Wuerzburg University Hospital
Other Study IDs: EA4/140/16
Record Dates: First submitted 2017-08-03; First posted 2017-08-11 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Stroke
Keywords: acute; informed consent; thrombolysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Patients with acute ischaemic stroke who were administered intavenous thrombolysis or patients with acute ischaemic stroke refusing intravenous thrombolysis; recall in both cases 60 to 90 minutes after the informed consent procedure
  Interventions: Other: Group 1
- Group 2: 1st of 2nd degree relatives of patients with acute ischaemic stroke, who witnessed the informed consent procedure
  Interventions: Other: Group 1
- Group 3: Stroke patients with acute or subacute ischaemic stroke with a contraindication for intravenous thrombolysis
  Interventions: Other: Group 1
- Group 4: Patients without an ischaemic stroke but similiar risk factors (admitted to the Departement of Cardiology and Pneumology, Charité, Campus Benjamin Franklin, Berlin, Germany)
  Interventions: Other: Group 1
- Group 5: Patients with acute ischaemic stroke who were administered intavenous thrombolysis - recall 24 hours after the informed consent procedure
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1
  Other Names: Group 2; Group 3; Group 4; Group 5

SUMMARY:
The aim of the study is to investigate the ability to recall information given during informed consent on intravenous thrombolysis in patients with acute ischaemic stroke.

DETAILED DESCRIPTION:
The purpose of this prospective multi-center study is to investigate whether patients with acute ischaemic stroke are able to recall information given before providing informed consent to intravenous thrombolysis after the end of treatment. Patients with acute ischaemic stroke will be compared to a group of relatives who witnessed the informed consent procedure of a relative with acute ischaemic stroke, stroke patients who were not treated with intravenous thrombolysis and patients without an ischaemic stroke but similiar risk factors (admitted to the Departement of Cardiology and Pneumology, Charité, Campus Benjamin Franklin, Berlin, Germany).

ELIGIBILITY:
Inclusion criteria (all):

* age ≥18 years
* able to give informed consent
* ability to understand and read German
* no prior i.v.-thrombolysis

Additional inclusion criteria - patients with acute ischaemic stroke:

* suspected ischaemic stroke (according to brain CT) or MRI-proven acute ischaemic stroke
* indication for intravenous thrombolysis

Additional inclusion criteria - relatives:

· relative (1st or 2nd dregree) of a patient with acute ischaemic stroke and present during the informed consent procedure

Additional inclusion criteria - stroke patients with a contraindication for thrombolysis:

* ischaemic stroke (according to brain MRI or CT)
* contraindication for intravenous thrombolysis

Additional inclusion criteria - non-stroke patients:

· present admission at the Department of Cardiology and Pneumology, Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, Germany

Exclusion criteria (all groups):

* not able to give imformed consent or under legal supervision/guardianship
* participation in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischaemic stroke and intravenous thrombolysis or patients with acute ischaemic stroke refusing intravenous thrombolysis, relatives (1st or 2nd degree) of patients with acute ischaemic stroke, patient with acute or subacute ischaemic stroke with a contraindication for intravenous thrombolysis and patients without acute ischaemic stroke (admitted to the Department of Cardiology (Charité, Campus Benjamin Franklin, Germany).
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Recall of the designated facts given during informed consent procedure on intravenous thrombolysis after acute ischaemic stroke | Within 24 hours

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Department of Neurology, University Hospital Würzburg, Würzburg, Bavaria
  - Department of Neurology, University Hospital Leipzig, Leipzig, Saxony
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Department of Neurology, University of Heidelberg, Heidelberg
  - Klinikum der Stadt Ludwigshafen a. Rh., Ludwigshafen am Rhein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuster L, Essig F, Daneshkhah N, Herm J, Hellwig S, Endres M, Dirnagl U, Hoffmann F, Michalski D, Pfeilschifter W, Urbanek C, Petzold GC, Rizos T, Kraft A, Haeusler KG. Ability of patients with acute ischemic stroke to recall given information on intravenous thrombolysis: Results of a prospective multicenter study. Eur Stroke J. 2023 Mar;8(1):241-250. doi: 10.1177/23969873221143856. Epub 2023 Jan 6. PMID 37021170